CLINICAL TRIAL: NCT05540340
Title: Pharmacokinetic Directed Melphalan for Lymphoma Patients Undergoing Autologous Hematopoietic Cell Transplantation
Brief Title: A Study of Melphalan in People With Lymphoma Getting an Autologous Hematopoietic Cell Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-086
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma; Lymphoma, B-Cell; Lymphoma, T-Cell; Lymphoma, Hodgkin; Lymphoma, Non-Hodgkin
Keywords: Pharmacokinetics; Carmustine; Etoposide; Melphalan; Cytarabine; 22-086
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Lymphoma, T-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Pharmacokinetic directed melphalan (Experimental): This is a feasibility study of pharmacokinetic (PK)-directed Captisol Enabled (CE) melphalan dosing to target an AUC of 8.5 (+/- 1.5) using a population PK model in lymphoma patients receiving BEAM [carmustine (BCNU) (B), etoposide (E), cytarabine (Ara-C) (A), and melphalan (M)], followed by autologous hematopoietic cell transplantation (AHCT). This study will enroll patients with lymphoma planned for BEAM-AHCT. Carmustine IV will be given on day -6, followed by etoposide IV and cytarabine IV from day -5 to -2 as per the MSK inpatient or outpatient standard of care. The calculated melphalan dose based on population PK model to achieve the proposed melphalan target exposure [8.5 (+/- 1.5) mg*h/L], will be administered on day -1, and six peripheral blood samples of 5 ml in lithium heparin tubes will be collected at 5, 15, 30, 40, 75, and 150 minutes after the melphalan, for PK testing to determine if the goal AUC was achieved.
  Interventions: Other: Pharmacokinetics
- Cohort 2: Pharmacokinetic directed melphalan (Experimental): In cohort 2, carmustine will be on Day -7, cytrabine and etoposide on Day -6 to Day -3, and melphalan (70mg/m2 /day IV) will be administered on day -2 followed by PK samples to determine the melphalan dose on day -1 using the population PK model. PK samples will be collected again after the dose on day -1 to confirm the total melphalan AUC of 8.5 (+/- 1.5) mg*h/L. Six peripheral blood samples of 5 ml in lithium heparin tubes will be collected at 5, 15, 30, 40, 75, and 150 minutes after the melphalan, for PK testing. The first four time points are +/- 2 min and the last two time points are +/- 5 minutes.
  Interventions: Other: Pharmacokinetics

INTERVENTIONS:
Other: Pharmacokinetics — Six peripheral blood samples of 5 ml in lithium heparin tubes will be collected at 5, 15, 30, 40, 75, and 150 minutes after the melphalan, for PK testing. The first four time points are +/- 2 min and the last two time points are +/- 5 minutes.
  Arms: Cohort 1: Pharmacokinetic directed melphalan
Other: Pharmacokinetics — Six peripheral blood samples of 5 ml in lithium heparin tubes will be collected at 5, 15, 30, 40, 75, and 150 minutes after the melphalan to determine the actual AUC achieved using the population PK.
  Arms: Cohort 2: Pharmacokinetic directed melphalan

SUMMARY:
The purpose of this study is to find out whether it is practical to use a newer way to calculate melphalan dose given (called population PK model) in BEAM chemotherapy before AHCT. Standard dose is fixed for everybody and is calculated using height and weight. The population PK model, tested in this study, uses information based on people who have previously received melphalan and aims to calculate an optimal dose separately for each person. Study researchers think that the dose calculated using the population PK model may still be effective but have less side effects than the standard melphalan dose.

ELIGIBILITY:
Inclusion Criteria:

* Age18 - 79 years old
* Diagnosed with any type of lymphoma [Hodgkin, non-Hodgkin (B- or T-cell)] and planned for BEAM-AHCT
* KPS > 70
* Cardiac ejection fraction of > 45%
* Hemoglobin-adjusted diffusing capacity of carbon monoxide (DLCO) of ≥45%
* Creatinine clearance of ≥ 40 mL/min
* Completion of most recent systemic therapy within 12 weeks of enrollment
* Complete or partial response to systemic chemotherapy by IWG Working Group Criteria.
* Total bilirubin < 2.0 mg/dL in the absence of suspected Gilbert's disease (if Gilbert's disease is suspected, the total bilirubin must be ≤3.0 mg/dL), and AST & ALT < 2.5 ULN.
* Minimum stem cell dose of 2 x 10*6 CD34+ cells/kg

Exclusion Criteria:

* Disease progression by IWG Working Group since last therapy
* Pregnant or lactating females
* Contraindication to CE melphalan or any of the required supportive treatments, including hypersensitivity to G-CSF or pegfilgrastim
* Any known allergy or allergic reactions to Captisol
* Any other medical condition or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
determine if this target AUC can be achieved | 1 year
  within a range of 8.5 (+/- 1.5) mg*h/L using population PK model.

CONTACTS AND LOCATIONS:
Overall Officials: Parastoo Dahi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm